CLINICAL TRIAL: NCT00963807
Title: Phase II Single-Arm Trial Comparing the Use of FLT PET to Standard Computed Tomography to Assess the Treatment Response of Neoadjuvant Docetaxel and Cisplatin in Stage IB-IIIA Resectable Non-small Cell Lung Cancer
Brief Title: A Comparison of FLT to FDG PET/CT in the Early Assessment of Chemotherapy Response in Stage IB-IIIA Resectable NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02899; NCI-2012-02899 (Other: CTRP (Clinical Trial Reporting Program)); NA_00017885 (Other: Johns Hopkins Medicine IRBs); J08134 (Other: JHU/Sidney Kimmel Comprehensive Cancer Center); NCI 8340 (Other: CTEP); N01CM00070 (NIH); P30CA006973 (NIH)
Record Dates: First submitted 2009-08-18; First posted 2009-08-24 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-01

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Fluorodeoxyglucose F18; alovudine; Magnetic Resonance Spectroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients receive docetaxel IV and cisplatin IV on day 1. Treatment repeats every 3 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo FDG PET/CT, FLT PET/CT, and thoracic CT at baseline and the end of cycles 1 and 2 and then undergo surgery.
  Interventions: Drug: Cisplatin; Procedure: CT; Drug: Docetaxel; Drug: FDG; Drug: FLT; Procedure: PET/CT; Procedure: Surgery

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: CT — Undergo FDG PET/CT, FLT PET/CT and thoracic CT
  Other Names: CAT; CAT Scan; Computed Tomography; Computerized Axial Tomography; Computerized Tomography; CT SCAN; tomography
Drug: Docetaxel — Given IV
  Other Names: RP56976; Taxotere; Taxotere Injection Concentrate
Drug: FDG — Undergo FDG PET/CT
  Other Names: 18FDG; fludeoxyglucose F 18; FLUDEOXYGLUCOSE F-18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: FLT — Undergo FLT PET/CT
  Other Names: 18F-FLT; 3'-deoxy-3'-(18F) fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; fluorothymidine F 18; FLUOROTHYMIDINE F-18
Procedure: PET/CT — Undergo FDG PET/CT and FLT PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Surgery — Undergo surgery
  Other Names: Therapeutic Conventional Surgery

SUMMARY:
This study is being done to compare a special type of Positron Emission Tomography (PET) scan with CT scan in patients with surgically removable lung cancer to see which method is more useful in measuring a response to treatment. A PET scan uses small amounts of radioactive material injected into the blood to show the internal workings of the body. In this study, we will use two radioactive materials: 18F-FLT (referred to as FLT) and 18F-FDG (referred to as FDG). FDG is used routinely in the staging of lung cancer and is approved by the FDA for that purpose. FLT is used in the special type of PET scan being assessed by this study. In addition the study will assess the effects of the combination of docetaxel and cisplatin (chemotherapeutic drugs) on certain pathological characteristics of the tumor. The combination of docetaxel and cisplatin is approved by the Food and Drug Administration (FDA) for the treatment of advanced/metastatic NSCLC (non-small cell lung cancer). It is not approved for use in patients who have surgically removable NSCLC. In such cases cisplatin is used as a single drug therapy before surgery. The FDA is allowing the use of docetaxel along with cisplatin in this research study.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the absolute decrease measured in primary tumor 18 F-F-3'-fluoro-3'-deoxy-L-thymidine (FLT) uptake (standard uptake value [SUV] and influx constant [Ki]) between pre-treatment imaging and imaging after the first cycle of therapy differs in patients categorized as responders or non-responders based on Response Evaluation Criteria in Solid Tumors (RECIST) measured with computed tomography (CT) after the second cycle of therapy.

SECONDARY OBJECTIVES:

I. To determine if the absolute decrease measured in primary tumor FDG uptake (SUV) between pre-treatment imaging and imaging after the first cycle of therapy differs in patients categorized as responders or non-responders based on RECIST measured with CT after the second cycle of therapy.

II. To assess the effects of the combination of docetaxel and cisplatin on fractional tumor viability and proliferative fraction pre and post treatment and to correlate these with the PET SUV data for both tracers.

III. To assess the methylation status of the checkpoint with forkhead and ring finger domains gene (CHFR) gene from pre-treatment tumor biopsies and correlate methylation status post treatment with clinical and pathologic response.

OUTLINE:

Patients receive docetaxel intravenously (IV) and cisplatin IV on day 1 and dexamethasone orally (PO) twice daily (BID). Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients undergo FDG PET/CT, FLT PET/CT, and thoracic CT at baseline and the end of courses 1 and 2 and then undergo surgery.

After completion of study treatment, patients are followed up for 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed clinical stage IB - IIIA non-small cell lung cancer; stage IV patients with oligometastatic disease with metastases that have been treated definitively with radiation or surgery are also eligible (ie: solitary brain or adrenal metastasis); mixed tumors will be categorized by the predominant cell type unless small cell elements are present in which case the patient is ineligible; note: tissue samples from biopsy confirmation will be required
* Patients must be surgically resectable as determined by a thoracic surgeon
* Patients must have measurable disease per RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with spiral CT scan
* Life expectancy of greater than 12 weeks
* ECOG performance status < 1
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 x institutional upper limit of normal
* AST (SGOT) =< 1.5 x institutional upper limit of normal
* Alkaline phosphatase =< 2.5 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/1.73 m2 for patients with creatinine levels above institutional normal
* Fasting screening blood glucose =< 200 mg/dL
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with either agent

Exclusion Criteria:

* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients may not be receiving any other investigational agents
* Patients must not have received prior systemic chemotherapy or radiation therapy for lung cancer; prior systemic chemotherapy or radiation for other malignancies over three years prior to study enrollment may be allowed at the discretion of the principal medical investigator
* Prior malignancy in the past 3 years, other than non-melanoma skin cancer and in situ carcinoma of the cervix
* Patients who report a hearing deficit at baseline, even if it does not require a hearing aid or intervention, or interfere with activities of daily life (Common Terminology Criteria for Adverse Events [CTCAE] grade 2 or higher)
* Peripheral neuropathy > CTCAE grade 1
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin, docetaxel, or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled diabetes, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric/social situations that would limit compliance with study requirements
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Inability to comply with study and/or follow-up procedures

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wahl, Principal Investigator — Johns Hopkins University Sidney Kimmel Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery): Patients receive docetaxel IV and cisplatin IV on day 1 and dexamethasone PO BID. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients undergo FDG PET/CT, FLT PET/CT, and thoracic CT at baseline and the end of courses 1 and 2 and then undergo surgery.
  Cisplatin: Given IV
  Computed Tomography: Undergo FDG PET/CT, FLT PET/CT and thoracic CT
  Dexamethasone: Given PO
  Docetaxel: Given IV
  Fludeoxyglucose F-18: Undergo FDG PET/CT
  Fluorothymidine F-18: Undergo FLT PET/CT
  Laboratory Biomarker Analysis: Correlative studies
  Positron Emission Tomography: Undergo FDG PET/CT and FLT PET/CT
  Therapeutic Conventional Surgery: Undergo surgery
Period: Overall Study
Arm/Group | Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery)
Started | 26
Completed Baseline Imaging | 11
Completed Post-Cycle 1 Imaging | 9
Completed Post-Cycle 2 FLT Imaging | 9
Completed Post-Cycle 2 FDG Imaging | 8
Completed | 8
Not Completed | 18
Not completed — Physician Decision | 2
Not completed — Reaction to study chemotherapy regimen | 1
Not completed — Disease progression | 15

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery)
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 56.4 [33 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in 18F-Fluorothymidine (FLT) Uptake
Description: Will be calculated by subtracting the uptake of the scan after the first cycle of chemotherapy from the uptake of the pre-treatment scan.. Change in FLT uptake will be measured using the maximum standard uptake value adjusted for lean body mass (SULmax), which is a measure of how much radiotracer (in this case FLT) is being consumed by cells.
Time Frame: Baseline and 3 weeks
Measure: Mean (Standard Deviation); unit: SULmax
Arm/Group | Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery)
Number analyzed (Participants) | 9
SULmax | -0.4 (1.9)

2. Primary Outcome: Change in FLT Uptake
Description: Will be calculated by subtracting the uptake of the scan after the second cycle of chemotherapy from the uptake of the pre-treatment scan.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: SULmax
Arm/Group | Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery)
Number analyzed (Participants) | 9
SULmax | 0.2 (3.8)

3. Primary Outcome: Change in FLT Uptake in Responders and Non-responders
Description: Unadjusted analysis will be performed utilizing students t-tests. If the data appears non-normal, the Wilcox on rank-sum test will be used rather than the t-test. Adjusted analysis will be performed utilizing logistic regression.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: SULmax
Groups:
- Responders: RECIST responders based on CT measurements performed after 2 cycles of neoadjuvant therapy.
- Non-Responders: RECIST non-responders based on CT measurements performed after 2 cycles of neoadjuvant therapy
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 3 | 6
SULmax | -1.8 (2.1) | 1.2 (4.1)
Statistical Analysis 1: Comparison: Responders vs Non-Responders; Test type: Superiority or Other; p = 0.336, t-test, 2 sided

4. Secondary Outcome: Change in 18F-Fluorodeoxyglucose (FDG) Uptake
Description: Will be calculated by subtracting the baseline FDG uptake from the post-cycle 2 uptake (as measured by SULmax).
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: SULmax
Arm/Group | Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery)
Number analyzed (Participants) | 8
SULmax | -3.8 (3.9)

5. Secondary Outcome: Overall Response Rate Reported as a Proportion of the Total Number of Patients Who Received at Least One Cycle of Therapy Assessed Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: RECIST version 1.1 was utilized for this outcome measure. A detailed description of RECIST 1.1 can be found here: Nishino M, Jackman DM, Hatabu H, Yeap BY, Cioffredi LA, Yap JT, et al. New Response Evaluation Criteria in Solid Tumors (RECIST) guidelines for advanced non-small cell lung cancer: comparison with original RECIST and impact on assessment of tumor response to targeted therapy. AJR Am J Roentgenol 2010;195:W221-8.
Time Frame: Up to 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery)
Number analyzed (Participants) | 9
percentage of participants | 33

ADVERSE EVENTS:
Arm/Group | Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery)
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Docetaxel, Cisplatin, Dexamethasone, and Surgery) (N=9)
Death (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenic Fever (Immune system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less